CLINICAL TRIAL: NCT02359799
Title: Home- and Lab-Based Passive and Active Movement Rehabilitation of Ankle Impairments in Children With Cerebral Palsy
Brief Title: Robotic Rehabilitation of Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00079369
Record Dates: First submitted 2015-01-26; First posted 2015-02-10 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Spastic Cerebral Palsy
Keywords: Cerebral palsy; Ankle Impairments; Robotic rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lab group (Experimental): Lab-based intervention includes 18 training sessions using the IntelliStretch in the lab .
  Interventions: Device: IntelliStretch
- Home group (Experimental): Home-based intervention includes 18 training sessions using the IntelliStretch at home.
  Interventions: Device: IntelliStretch

INTERVENTIONS:
Device: IntelliStretch — The impaired ankle of the participants are trained 3 times a week for 6 weeks in the lab or at home. The participants use the portable robotic device to stretch the ankle and increase range of motion (ROM). Then subjects use their gained ROM immediately in the active movement training to play video games and improve motor control.

SUMMARY:
The purpose of the study is to examine the outcomes of home-based robot-guided therapy and compare it to laboratory-based robot-guided therapy for impaired ankles in cerebral palsy. Children with spastic cerebral palsy (CP) are randomly placed into two groups, participating in robot-guided stretching and active movement training either in a research lab setting (Lab group) or in a home setting (Home group).

DETAILED DESCRIPTION:
Children with spastic CP will be randomly placed to 2 groups, either a Lab group or a Home group. For both groups, the participation will involve 18 training sessions over 6 weeks with 3 sessions each week. Each training session will last about 45 minutes, including stretching and active movement training.

The participant will be asked to sit with the foot secured to a footplate and leg fixed by a leg-support. Once the rehab robot is on the child's ankle, the investigator will first determine maximum range of motion that is safe for the ankle stretching. The robot will then move the ankle joint slowly within the set range of motion, and stretch the ankle back and forth. The passive stretching will help loosen the child's muscle and increase range of motion in the ankle joint. Passive stretching will last about 15 minutes.

After stretching, the investigator will ask the child to move and control the ankle joint back and forth to complete video-game tasks. While the child moves the ankle, the robot will provide assistance or resistance to improve control of the ankle joint. Active movement training will last about 20 minutes.

For Home group, the family members will be trained by the research team at the lab on how they use the rehab robot properly. On the day of the first assessment, the investigator will go through the device operation with family members. A detailed user manual will be given. The investigator will allow the family members and the child to practice using the device as many times as needed until the participant feel comfortable using the device at home. The family members should prepare for a minimum of one hour for this instructional period to learn the device, but they will be allowed as much time as needed.

Before leaving UMB to begin at-home training, the family members will be checked for the competency of using the device. The family members will be asked to go through each step without any direct assistance with the research staff. The family members may use their own vehicle to take the portable rehab robot home. While the family members are doing training for the child at home, the training data will be saved automatically in the laptop with the rehab robot.

Only one ankle joint will be allowed to treat using this robotic device. The investigator will choose the more impaired side ankle of the child to start the training. The investigator will follow up with the family members 1-3 times per week to check in regarding the child's participation and any issues during the training. The family members can also call the research staff if they have any questions about the training. The family members should follow the same training plan during 18 training sessions unless the investigator decide to adjust the training setups based on the child's progress.

Outcome assessments

During the study, the child will have 3 assessment visits in the research lab. The visits will occur before and after 6-week training, and at a follow-up 6 weeks after the training ends. During the assessment, the child's ankle will be moved by the robot to test passive range of motion and joint stiffness. The participant will also move the ankle himself and the active range of motion and muscle strength will be recorded. Clinical exam scales will be done including modified Ashworth scale, Selective Control Assessment of Lower Extremity (SCALE), balance, and walking ability (distance covered in 6 minutes).

ELIGIBILITY:
Inclusion Criteria:

1. Spastic cerebral palsy with diplegia or hemiplegia (affected both legs or one leg)
2. 6-17 years old
3. Can follow instructions and express any discomfort during the sessions.

Exclusion Criteria:

1. Orthopedic surgery, serial casting, or injection of muscle relaxants such as botulinum toxin type A within 6 months prior to participation in the study
2. Severe ankle contracture, greater than 20° plantar flexion
3. Other unrelated neurological impairments or musculoskeletal injuries
4. Can not sit for 1 hour

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Changes of Active Range of Motion (AROM) | AROM will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  The subjects will be asked to use their muscles to move the ankle joint and record the range of motion by the robot.

SECONDARY OUTCOMES:
Changes of Modified Ashworth Scale (MAS) | MAS will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  The MAS measures spasticity in patients with lesions of the Central Nervous System.
Changes of Selective Control Assessment of Lower Extremity (SCALE) | SCALE will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  SCALE is a clinical assessment developed to quantify selective voluntary motor control in patients with cerebral palsy
Changes of Pediatric Balance Scale (PBS) | PBS will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  PBS is a 14-item criterion-referenced measure that examines functional balance in the context of everyday tasks in the pediatric population.
Changes of the Timed Up and Go Test (TUG) | TUG will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  TUG assesses mobility, balance, walking ability, and fall risk.
Changes of 6 Minute Walk Test (6MWT) | 6MWT will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  The test assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
Changes of Passive Range of Motion (PROM) | PROM will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  The robot will move the ankle joint of the subjects and record the range of motion.
Changes of the muscle strength | The muscle strength will be assessed at 3 time points: at the beginning and the end of 6-week training, and follow-up at 6 weeks after the training ends.
  Dorsiflexor and plantarflexor strength will be measured with the ankle keeping held at 0° dorsiflexion.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Zhang, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engsberg JR, Ross SA, Olree KS, Park TS. Ankle spasticity and strength in children with spastic diplegic cerebral palsy. Dev Med Child Neurol. 2000 Jan;42(1):42-7. doi: 10.1017/s0012162200000086. PMID 10665974
- [Background] Krebs HI, Hogan N, Aisen ML, Volpe BT. Robot-aided neurorehabilitation. IEEE Trans Rehabil Eng. 1998 Mar;6(1):75-87. doi: 10.1109/86.662623. PMID 9535526
- [Background] Damiano DL, Alter KE, Chambers H. New clinical and research trends in lower extremity management for ambulatory children with cerebral palsy. Phys Med Rehabil Clin N Am. 2009 Aug;20(3):469-91. doi: 10.1016/j.pmr.2009.04.005. PMID 19643348
- [Background] Novak I, McIntyre S, Morgan C, Campbell L, Dark L, Morton N, Stumbles E, Wilson SA, Goldsmith S. A systematic review of interventions for children with cerebral palsy: state of the evidence. Dev Med Child Neurol. 2013 Oct;55(10):885-910. doi: 10.1111/dmcn.12246. Epub 2013 Aug 21. PMID 23962350
- [Background] Zhang M, Davies TC, Xie S. Effectiveness of robot-assisted therapy on ankle rehabilitation--a systematic review. J Neuroeng Rehabil. 2013 Mar 21;10:30. doi: 10.1186/1743-0003-10-30. PMID 23517734
- [Background] Selles RW, Li X, Lin F, Chung SG, Roth EJ, Zhang LQ. Feedback-controlled and programmed stretching of the ankle plantarflexors and dorsiflexors in stroke: effects of a 4-week intervention program. Arch Phys Med Rehabil. 2005 Dec;86(12):2330-6. doi: 10.1016/j.apmr.2005.07.305. PMID 16344031
- [Background] Wu YN, Hwang M, Ren Y, Gaebler-Spira D, Zhang LQ. Combined passive stretching and active movement rehabilitation of lower-limb impairments in children with cerebral palsy using a portable robot. Neurorehabil Neural Repair. 2011 May;25(4):378-85. doi: 10.1177/1545968310388666. Epub 2011 Feb 22. PMID 21343525
- [Background] Willerslev-Olsen M, Andersen JB, Sinkjaer T, Nielsen JB. Sensory feedback to ankle plantar flexors is not exaggerated during gait in spastic hemiplegic children with cerebral palsy. J Neurophysiol. 2014 Feb;111(4):746-54. doi: 10.1152/jn.00372.2013. Epub 2013 Nov 13. PMID 24225545
- [Background] Geiger R, Strasak A, Treml B, Gasser K, Kleinsasser A, Fischer V, Geiger H, Loeckinger A, Stein JI. Six-minute walk test in children and adolescents. J Pediatr. 2007 Apr;150(4):395-9, 399.e1-2. doi: 10.1016/j.jpeds.2006.12.052. PMID 17382117
- [Background] Ballaz L, Plamondon S, Lemay M. Ankle range of motion is key to gait efficiency in adolescents with cerebral palsy. Clin Biomech (Bristol). 2010 Nov;25(9):944-8. doi: 10.1016/j.clinbiomech.2010.06.011. Epub 2010 Jul 23. PMID 20655641
- [Background] Gao F, Ren Y, Roth EJ, Harvey R, Zhang LQ. Effects of repeated ankle stretching on calf muscle-tendon and ankle biomechanical properties in stroke survivors. Clin Biomech (Bristol). 2011 Jun;26(5):516-22. doi: 10.1016/j.clinbiomech.2010.12.003. Epub 2011 Jan 6. PMID 21211873
- [Background] Mankodi A, Azzabou N, Bulea T, Reyngoudt H, Shimellis H, Ren Y, Kim E, Fischbeck KH, Carlier PG. Skeletal muscle water T2 as a biomarker of disease status and exercise effects in patients with Duchenne muscular dystrophy. Neuromuscul Disord. 2017 Aug;27(8):705-714. doi: 10.1016/j.nmd.2017.04.008. Epub 2017 Apr 28. PMID 28601553
- [Background] Sukal-Moulton T, Clancy T, Zhang LQ, Gaebler-Spira D. Clinical application of a robotic ankle training program for cerebral palsy compared to the research laboratory application: does it translate to practice? Arch Phys Med Rehabil. 2014 Aug;95(8):1433-40. doi: 10.1016/j.apmr.2014.04.010. Epub 2014 May 2. PMID 24792141
- [Derived] Chiu HC, Ada L, Bania TA. Mechanically assisted walking training for walking, participation, and quality of life in children with cerebral palsy. Cochrane Database Syst Rev. 2020 Nov 18;11(11):CD013114. doi: 10.1002/14651858.CD013114.pub2. PMID 33202482
- [Derived] Chen K, Wu YN, Ren Y, Liu L, Gaebler-Spira D, Tankard K, Lee J, Song W, Wang M, Zhang LQ. Home-Based Versus Laboratory-Based Robotic Ankle Training for Children With Cerebral Palsy: A Pilot Randomized Comparative Trial. Arch Phys Med Rehabil. 2016 Aug;97(8):1237-43. doi: 10.1016/j.apmr.2016.01.029. Epub 2016 Feb 20. PMID 26903143